CLINICAL TRIAL: NCT06554041
Title: Soft Tissue Response to Different Restorative Materials Used in Implant Dentistry
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Harvard Medical School (HMS and HSDM) (Other)
Responsible Party: Principal Investigator, Samuel Akhondi, Research Associate, Harvard Medical School (HMS and HSDM)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: BE-2-106
Record Dates: First submitted 2024-08-05; First posted 2024-08-14 (Actual); Last update posted 2024-08-14 (Actual); Status verified 2024-08

CONDITIONS: Edentulous Alveolar Ridge; Peri-Implantitis; Peri-implant Mucositis; Prosthetic Infection; Prosthetic Complication
Keywords: Dental Implants; Peri-Implant Soft Tissue; Prosthetic Materials; Inflammation Markers; Oral Health
MeSH Terms: conditions — Peri-Implantitis | interventions — Crowns

STUDY DESIGN:
Intervention Model Description: This clinical trial employs an interventional study model with a parallel assignment. A total of 40 edentulous patients, will be randomized into four groups.
  The study is open-label, meaning that both the researchers and the participants will know which material is being used for each patient. This design is intended to evaluate the impact of these different materials on the health of the peri-implant soft tissue by measuring inflammatory markers and clinical outcomes such as bleeding on probing and pocket depth over a six-month period.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Dental Crown with Titanium-Abutment (Experimental): Participants in this arm will receive dental implants and single crowns made from titanium. The impact of titanium on peri-implant soft tissue health will be evaluated by measuring inflammatory markers and clinical outcomes such as bleeding on probing and pocket depth at 3 and 6 months post-implantation.
  Interventions: Device: Dental Crown with Titanium-Abutment
- Dental Crown with PEEK (Polyetheretherketone)-Abutment (Experimental): Participants in this arm will receive dental implants and single crowns made from PEEK. The study will assess the biocompatibility of PEEK by examining inflammatory responses and clinical outcomes, including bleeding on probing and pocket depth, at 3 and 6 months post-implantation.
  Interventions: Device: Dental Crown with PEEK (Polyetheretherketone)-Abutment
- Dental Crown with Zirconia-Abutment (Experimental): Participants in this arm will receive dental implants and single crowns made from zirconia. The effects of zirconia on peri-implant soft tissue will be analyzed by measuring the levels of inflammatory markers and observing clinical outcomes such as bleeding on probing and pocket depth at 3 and 6 months post-implantation.
  Interventions: Device: Dental Crown with Zirconia-Abutment
- Dental Crown with Lithium-Disilicate-Abutment (e.max) (Experimental): Participants in this arm will receive dental implants and single crowns made from lithium disilicate (e.max). The study will evaluate the biocompatibility of e.max by measuring inflammatory markers and clinical outcomes, including bleeding on probing and pocket depth, at 3 and 6 months post-implantation.
  Interventions: Device: Dental Crown with Lithium-Disilicate-Abutment (e.max)

INTERVENTIONS:
Device: Dental Crown with Titanium-Abutment — Participants in this clinical trial will receive dental implants and single screw-retained crowns made from one of four different materials: titanium, PEEK (Polyetheretherketone), zirconia, or lithium disilicate (e.max). The implants will be placed in the posterior region of the mandible or maxillae. The study will evaluate the impact of these materials on peri-implant soft tissue health by measuring inflammatory markers in the peri-implant crevicular fluid and assessing clinical outcomes such as bleeding on probing and pocket depth at 3 and 6 months post-implantation.
  Arms: Dental Crown with Titanium-Abutment
Device: Dental Crown with PEEK (Polyetheretherketone)-Abutment — Participants in this clinical trial will receive dental implants and single screw-retained crowns made from one of four different materials: titanium, PEEK (Polyetheretherketone), zirconia, or lithium disilicate (e.max). The implants will be placed in the posterior region of the mandible or maxillae. The study will evaluate the impact of these materials on peri-implant soft tissue health by measuring inflammatory markers in the peri-implant crevicular fluid and assessing clinical outcomes such as bleeding on probing and pocket depth at 3 and 6 months post-implantation.
  Arms: Dental Crown with PEEK (Polyetheretherketone)-Abutment
Device: Dental Crown with Zirconia-Abutment — Participants in this clinical trial will receive dental implants and single screw-retained crowns made from one of four different materials: titanium, PEEK (Polyetheretherketone), zirconia, or lithium disilicate (e.max). The implants will be placed in the posterior region of the mandible or maxillae. The study will evaluate the impact of these materials on peri-implant soft tissue health by measuring inflammatory markers in the peri-implant crevicular fluid and assessing clinical outcomes such as bleeding on probing and pocket depth at 3 and 6 months post-implantation.
  Arms: Dental Crown with Zirconia-Abutment
Device: Dental Crown with Lithium-Disilicate-Abutment (e.max) — Participants in this clinical trial will receive dental implants and single screw-retained crowns made from one of four different materials: titanium, PEEK (Polyetheretherketone), zirconia, or lithium disilicate (e.max). The implants will be placed in the posterior region of the mandible or maxillae. The study will evaluate the impact of these materials on peri-implant soft tissue health by measuring inflammatory markers in the peri-implant crevicular fluid and assessing clinical outcomes such as bleeding on probing and pocket depth at 3 and 6 months post-implantation.
  Arms: Dental Crown with Lithium-Disilicate-Abutment (e.max)

SUMMARY:
The goal of this clinical trial is to learn how different materials used in dental implants affect the surrounding gum tissue in adults who need dental implants. The main questions it aims to answer are:

How do different materials (titanium, PEEK, zirconia, and lithium disilicate) affect inflammation around dental implants? What changes occur in inflammation markers in the gum tissue after 3 and 6 months? Researchers will compare the different materials to see which one causes the least amount of inflammation.

Participants will:

Receive dental implants made from different materials. Have samples of fluid from around their implants collected for analysis at 3 and 6 months.

Undergo regular dental check-ups to measure gum health, such as bleeding and pocket depth around the implants.

DETAILED DESCRIPTION:
The study will involve a total of 40 edentulous patients, each missing four teeth in the posterior region of the mandible or maxillae. Each patient will receive four dental implants and single crowns made from different materials. The primary objectives are to evaluate biomarkers in peri-implant crevicular fluid and to assess the changes in these biomarkers after three and six months of loading. This research will help determine the biocompatibility of the materials and their potential to cause peri-implantitis.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be 18 years or older.
* Participants must be edentulous with at least four missing teeth in the posterior region of the mandible or maxillae.
* Participants must have appropriate oral hygiene and periodontal status of natural teeth, with a pocket depth of 4mm or less and no bleeding.
* Dental implants must be fully integrated with no bone resorption or inflammation after three months of implant placement, confirmed by X-ray and clinical examination.
* Implant placement must be into natural bone without additional procedures such as sinus lift or bone augmentation.
* The procedure must be a standard implantation with no immediate implant placement.
* The height of the gingiva must be at least 3mm or more.

Exclusion Criteria:

* Patients with systemic diseases such as malignancy, diabetes, osteoporosis, or rheumatoid arthritis.
* Patients with a history of periodontal treatment.
* Patients who smoke or use tobacco.
* Patients who have received antibiotic treatment within three months prior to implantation.
* Pregnant individuals.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-08-23 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Concentration of Inflammatory Biomarkers in Peri-Implant Crevicular Fluid | 3 and 6 months post-implantation
  The primary outcome measure will evaluate the concentration of inflammatory biomarkers in the peri-implant crevicular fluid, including IL-6, IL-8, IL-10, IL-17, TNF-alpha, IL-12, IL-1-beta, and IL-4. These biomarkers all have the same unit and will be measured to assess the inflammatory response of peri-implant soft tissue to different prosthetic materials (titanium, PEEK, zirconia, and lithium disilicate). The goal is to determine which material induces the least amount of inflammation, indicating better biocompatibility and a lower risk of peri-implantitis.

SECONDARY OUTCOMES:
Clinical Measurements of Bleeding on Probing (BOP) and Pocket Depth | 3 and 6 months post-implantation
  The secondary outcome measure will assess the clinical health of the peri-implant tissue by measuring bleeding on probing (BOP) around the dental implants. These clinical parameters will provide additional insights into the soft tissue response to the different prosthetic materials used in the implants (titanium, PEEK, zirconia, and lithium disilicate). Improved clinical outcomes, such as reduced bleeding and shallower pocket depths, will indicate better biocompatibility and integration of the implant materials.
Clinical Measurements of Pocket Depth | 3 and 6 months post-implantation
  The secondary outcome measure will assess the clinical health of the peri-implant tissue by measuring pocket depth around the dental implants. These clinical parameter will provide additional insights into the soft tissue response to the different prosthetic materials used in the implants (titanium, PEEK, zirconia, and lithium disilicate). Improved clinical outcomes, such as reduced bleeding and shallower pocket depths, will indicate better biocompatibility and integration of the implant materials.

CONTACTS AND LOCATIONS:
Locations (1):
- VIC Clinic, Vilnius, Lithuania

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) will be made available to other researchers upon reasonable request. The data will include de-identified participant data, relevant clinical and biochemical measurements, and any other pertinent data collected during the study.
Supporting Information: Study Protocol
Time Frame: Data will be available after the primary and secondary outcomes have been published, and will remain accessible for five years following the end of the study.
Access Criteria: Researchers can request access to the IPD by contacting the principal investigator. Requests should include a research proposal and a data use agreement.